CLINICAL TRIAL: NCT06284642
Title: Effectiveness and Safety of Early Lumbar Drainage Combined With Intrathecal Urokinase Injection in the Treatment of Severe Aneurysmal Subarachnoid Hemorrhage (LD-ITUK): a Multicentral Randomized Control Trial
Brief Title: Early Lumbar Drainage Combined With Intrathecal Urokinase Injection for Treatment of Severe Aneurysmal SAH (LD-ITUK)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LD-ITUK-2024-001
Record Dates: First submitted 2024-02-01; First posted 2024-02-29 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-12

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Urokinase-Type Plasminogen Activator; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lumbar drainage combined with intrathecal urokinase injection (Active Comparator): lumbar drainage combined with intrathecal urokinase injection
  Interventions: Drug: Urokinase
- lumbar drainage (Placebo Comparator): lumbar drainage combined with intrathecal placebo saline injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Urokinase — On the basis of standard treatment for severe neurological conditions, within 24 hours of aneurysm treatment, lumbar drainage combined with intrathecal urokinase injection was started. 30,000 IU urokinase dissolved in 3 ml normal saline was injected into the subarachnoid space, 3 ml normal saline was rinsed into the tube, and the tube was clamped for observation for 2 hours, once a day, for 3 consecutive days. Lumbar cisternae drainage Cerebrospinal fluid is slowly and steadily drained at a rate of less than 8ml/h per hour, the daily drainage volume is not more than 200 ml, and the drainage time of lumbar cisternae is controlled within 7 to 10 days, not more than 14 days.
  Other Names: Urokinase-type plasminogen activator
  Arms: lumbar drainage combined with intrathecal urokinase injection
Drug: Placebo — On the basis of standard treatment for severe neurological conditions, the treatment of lumbar drainage combined with intrathecal placebo saline injection was started within 24 hours after aneurysm treatment, 3 ml placebo was injected into the subarachnoid space, 3 ml normal saline was flushed into the tube, and the tube was observed for 2 hours, once a day for 3 consecutive days. Lumbar cisternae drainage Cerebrospinal fluid is slowly and steadily drained at a rate of less than 8ml/h per hour, the daily drainage volume is not more than 200 ml, and the drainage time of lumbar cisternae is controlled within 7 to 10 days, not more than 14 days.
  Other Names: Saline
  Arms: lumbar drainage

SUMMARY:
The LD-ITUK is a multicenter, prospective, randomized, double-blind, blind endpoint, placebo-control design trial. All eligible patients with the diagnosis of severe aSAH will be randomly assigned to the treatment group or the placebo group. Patients in the treatment group will receive standard treatment with the addition of lumbar drainage combined with intrathecal urokinase injection started within 24 hours after aneurysm treatment with 30000 IU urokinase, once a day for 3 consecutive days. Patients in the control group will receive standard treatment with the addition of lumbar drainage combined with intrathecal placebo (0.9%NaCl) injection. The primary outcome measure is favorable functional outcome, defined as a score of 0 to 2 on the modified Rankin Scale (mRS), at 6 months after aneurysmal SAH. Primary outcome will be determined by a member of the Independent Committee on Terminal events.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhages (aSAH) represent about 8% of all strokes and 9.8 per 100,000 per year in China, which is higher than the overall annual incidence rate worldwide. The cumulative death rate after-onset represent about 24.6% in China, only about 30% survivors will be able to have a good neurological prognosis, the majority of the remaining survivors suffer from long-term disability or cognitive impairment. However, these condition may be even worse in patients with severe aSAH.

Studies suggest that early clearance of subarachnoid clot may be associated with a good neurological prognosis. Indeed, subarachnoid clot aggravate the phenomena of cerebral vasospasm and delayed cerebral ischemia in the delayed phase, and promote cell injure within the hypoperfusion zone of the brain in the longer term. Thus, early removal of subarachnoid clot may have a favorable effect on neurological prognosis. Current aSAH recommendations and guidelines advocate the use of lumbar drainage only in case of acute hydrocephalus. The EARLYDRAIN trial suggests that lumber cerebrospinal fluid drainage can early remove subarachnoid clot compare to the standard neurocritical treatment, and improve the prognosis after aSAH. However, the ratio of unfavorable prognosis in severe aSAH is still high.

Intrathecal urokinase injection has been proved to effeciently remove the subarachnoid clot, however, no randomized control trials have been conducted to evaluate the improvement of lumbar drainage combined with intrathecal urokinase injection in the favorable functional outcome, defined as a score of 0 to 2 on the modified Rankin Scale (mRS), at 6 months after aneurysmal SAH.

The LD-ITUK trial was designed to evaluate whether severe aSAH treated by standard treatment with the addition of lumbar drainage combined with intrathecal urokinase injection have a significantly higher percentage of favourable outcome after six months (score 0-2 on the Modified Rankin Scale) compared to the placebo treated by standard treatment with the addition of lumbar drainage combined with intrathecal placebo (0.9%NaCl) injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age ≥ 18 years
* First occurrence of aneurysmal subarachnoid hemorrhage
* Patients without any craniotomy treatment before onset
* Hunt-Hess grade III-V
* mRS grade 0 or 1 before onset
* Aneurysm treatment within 48 hours of onset
* Informed consent given by the subject or guardian

Exclusion Criteria:

* Subarachnoid hemorrhage caused by arteriovenous malformation or moyamoya disease or other cerebrovascular disease
* Patients requiring craniotomy to remove intracranial hematoma
* modified Fisher Scale grade 0
* Prothrombin time (PT) and activated partial thromboplastin time (APTT) are greater than 2 times the extended range
* Absolute contraindications for lumbar puncture (e.g., brain hernia, puncture site infection)
* Patients with a life expectancy of less than 1 year due to other causes
* Other concomitant serious diseases that are difficult to treat;
* Pregnant woman
* Patients who were known to be allergic to urokinase and excipients or had a history of severe allergy and were deemed unsuitable for inclusion by the investigators
* Participated in another interventional clinical trial within 30 days before randomization
* Other reasons deemed unsuitable for study participation by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 180 days
  Good (mRS 0-2) and Poor (mRS 3-6)

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  Good (mRS 0-2) and Poor (mRS 3-6)
Relative Modified Rankin Scale (mRS) | 90 days, 180 days
  Good (mRS 0-3) and Poor (mRS 4-6)
Modified Rankin Scale (mRS) distribution | 180 days
  On the distributed proportion in scores (0-6) on the mRS
Glasgow Outcome Scale (GOS） | 180 days
  Good (GOS 4-5) and Poor (GOS 1-3)
Questionnaire EuroQol Five Dimensions Questionnaire (EQ-5D) | 180 days
  EQ-5D questionnaires have 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 3 problem levels corresponding to patient response choices.
Barthel Index for Activities of Daily Living (BI) | 180 days
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.
Total hospitalized time | Discharge (assessed up to 30 days)
  Toal hospitalized time from ofter-onset to discharge, including neurocritical care unit
Total hospitalized costs | Discharge (assessed up to 30 days)
  Toal hospitalized costs from ofter-onset to discharge
Cerebral vasospasm (CV) | 14 days
  Occurence of any symptomatic or image CV after aSAH
Delayed cerebral ischemia (DCI) | 14 days
  Occurence of any symptomatic or image DCI after aSAH
Death | 180 days
  Occurence of any death during follow-up after operation
Hydrocephalus | 180 days
  Occurence of a hydrocephalus after-onset
Rebleeding | 30 days
  Occurence of a rebleeding after-onset

OTHER OUTCOMES:
Subarachnoid hemorrhage volume clearance | 30 days
  dynamic clearance of subarachnoid hemorrhage volume on non-contrast CT scans ofter-onset to discharge
Correlationship between cerebralspinal fluid pressure with subarachnoid hemorrhage volume | 72 hours after-onset
  correlationship between admission cerebralspinal fluid pressure with subarachnoid hemorrhage volume
Correlationship between clinical grades and subarachnoid hemorrhage volume | 72 hours after-onset
  correlationship between Hunt-Hess grade, WFNS, modified Fisher scale with subarachnoid hemorrhage volume

CONTACTS AND LOCATIONS:
Overall Officials: Xingen Zhu, MS, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No